CLINICAL TRIAL: NCT06261957
Title: A Randomized, Double-blind, Parallel Group, Multi-center Study to Evaluate the Long-term Safety of Salbutamol Rescue Medication When Administered Via Metered Dose Inhalers Containing the Propellant HFA-152a or Reference HFA-134a
Brief Title: A Study to Assess and Compare Safety and Tolerability of 3 Months Treatment With Salbutamol Administered Via MDI Containing Propellant HFA-152a or HFA-134a in Participants ≥ 18 Years of Age With Asthma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 220735; 2023-509001-76-00 (Other: EU CT Number)
Record Dates: First submitted 2024-02-08; First posted 2024-02-15 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Asthma
Keywords: Asthma; Salbutamol; MDI; HFA-152a; HFA-134a
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Salbutamol Test Arm (Experimental)
  Interventions: Drug: Salbutamol HFA-152a
- Salbutamol Reference Arm (Active Comparator)
  Interventions: Drug: Salbutamol HFA-134a

INTERVENTIONS:
Drug: Salbutamol HFA-134a — 100 microgram (μg) (ex-valve) at 30-second intervals per actuation
  Arms: Salbutamol Reference Arm
Drug: Salbutamol HFA-152a — 100 μg (ex-valve) at 30-second intervals per actuation
  Arms: Salbutamol Test Arm

SUMMARY:
The goal of this study is to assess and compare the safety and tolerability of salbutamol administered via metered dose inhaler (MDI) containing propellant 1,1-difluoroethane (HFA-152a) or 1,1,1,2-tetrafluoroethane (HFA-134a) in participants aged >=18 years with asthma

ELIGIBILITY:
Inclusion Criteria:

1. Participant of ≥18 years of age at the time of signing the informed consent or written informed consent is obtained from each study participant's legal guardian.
2. Asthma for ≥ 6 months, defined as:

   * Documented history of asthma, as defined by Global Initiative for Asthma (GINA) (GINA, 2023]
   * Receiving one of the following asthma treatments, at a stable dose (applicable to daily Inhaled corticosteroid (ICS), ICS/Long-acting bronchodilator (LABA), and ICS/LABA/Long-acting muscarinic antagonist [LAMA]), for at least 12 weeks prior to the screening visit, with treatment that is anticipated to remain stable for the duration of the study:

     * Short-Acting Beta-2-Adrenoreceptor Agonists (SABA) used as needed for asthma symptoms
     * Daily maintenance low to medium dose Inhaled corticosteroid (ICS) (low to medium dose ICS defined as 100-500 μg/day fluticasone propionate or equivalent as defined in the 2023 GINA guidelines [GINA, 2023], plus Short-Acting Beta-2-Adrenoreceptor Agonists (SABA), which is anticipated to remain stable for the duration of the study.
     * Daily maintenance low to medium dose ICS/ Long-acting bronchodilator (LABA) (low to medium dose ICS defined as 100-500 μg/day fluticasone propionate or equivalent as defined in the GINA guidelines [GINA, 2023] plus SABA, which is anticipated to remain stable for the duration of the study.
     * Daily maintenance ICS/LABA/LAMA (low to medium dose ICS defined as 100-500 µg/day fluticasone propionate or equivalent as defined in the GINA guidelines [GINA, 2023] plus SABA, which is anticipated to remain stable for the duration of the study.
     * Participants who utilize combination budesonide/formoterol as reliever therapy, whether or not this is in addition to a SABA - are not eligible for screening.
     * Participants who utilize ICS/SABA combination therapy as reliever therapy, in addition to low to medium dose ICS or ICS/LABA as maintenance, are only eligible if they agree to discontinue their ICS/SABA inhaler for the duration of the study (screening through follow-up).
3. Severity of disease assessed by the investigator by baseline pre-bronchodilator Forced expiratory volume in 1 second (FEV1)
4. Asthma Control Status

   * Asthma Control Questionnaire (ACQ) 6 score <1.5 at screening
   * Asthma that has remained stable with no severe exacerbations in the last 6 months. Severe exacerbation defined as:

     * Deterioration of asthma-requiring the use of systemic corticosteroids (tablets, suspension or injection), for at least 3 days, OR
     * An inpatient hospitalization or Emergency Department (ED) visit because of asthma, requiring systemic corticosteroids.
5. Evidence of reversibility of disease: Airway reversibility is defined as ≥12 percent (%) and ≥200 milliliter (mL) increase in FEV1 within 20 to 60 minutes following up to 4 inhalations of albuterol/salbutamol aerosol.
6. Participants on as-needed SABA only, or daily maintenance ICS (plus as needed SABA):

   * With a documented history of reversibility (as defined above) within 2 years will meet this inclusion criterion. Pre- and post-bronchodilator measurements will still be collected at screening to characterize the degree of reversibility.
   * Who do not have a documented history of reversibility within the past 2 years will need to demonstrate reversibility during the screening period.

     * SABA should be withheld for ≥6 hours
     * Participants on daily maintenance ICS/LABA or ICS/LABA/LAMA:
7. Participants on daily maintenance ICS/LABA or ICS/LABA/LAMA:

   * Do not need to demonstrate reversibility in accordance with the above definition during the screening period. A reversibility maneuver will be performed to characterize the degree of post-bronchodilator change.

     * SABA should be withheld for ≥6 hours
     * LABA- and LAMA-containing medications should be withheld for >=24 hours for the characterization of post-bronchodilator change.

Participants should be able to withhold SABA for ≥6 hours and LABA-/ LAMA containing medications for ≥24 hours for the purposes of performing screening spirometry.

Exclusion Criteria:

1. A history of life-threatening asthma or asthma that is unstable in the opinion of the investigator.
2. Other significant pulmonary diseases to include (but not limited to): pneumothorax, pulmonary fibrotic disease, bronchopulmonary dysplasia, chronic bronchitis, emphysema, chronic obstructive pulmonary disease, tuberculosis or other respiratory abnormalities other than asthma.
3. Respiratory Infection: Culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear that is not resolved within 4 weeks of screening that led to a change in asthma management, OR in the opinion of the Investigator, is expected to affect the participant's asthma status, OR the participant's ability to participate in the study.
4. Asthma Exacerbation: Any severe asthma exacerbation within 6 months prior to screening.
5. Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones) Biologic/immunosuppressive therapies used for the treatment of respiratory diseases during the 6 months, or 5 half-lives-whichever is longer-prior to start of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2025-09-05 (Estimated); Study Completion 2025-09-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to 3 months

SECONDARY OUTCOMES:
Number of participants with Serious Adverse Events (SAEs) | Up to 3 months
Absolute Values of Minimum serum potassium (milliequivalents per litre [mEq/L]) | Up to 3 months
Absolute values of serum potassium (milligrams per decilitre) | Up to 3 months
Change from baseline in serum potassium (milligrams per decilitre) | Baseline (Day 1) and up to 3 months
Absolute value of haematology parameter: Platelet count (cells per microliter) | Up to 3 months
Absolute value of haematology parameter: Red Blood Cell Count (RBC) (million cells per microliter) | Up to 3 months
Absolute value of haematology parameter: Mean Corpuscle Volume (MCV) (Femtoliters) | Up to 3 months
Absolute value of haematology parameter: Mean Corpuscle haemoglobin (MCH) (Picograms) | Up to 3 months
Absolute values of haematology parameter: Reticulocytes (Percentage of reticulocytes) | Up to 3 months
Absolute values of haematology parameters: Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils (giga cells per litre) | Up to 3 months
Absolute values of haematology parameter: haemoglobin (Hgb) (grams per decilitre) | Up to 3 months
Absolute values of haematology parameter: haematocrit (Proportion of red blood cells in blood) | Up to 3 months
Absolute values of Clinical Chemistry parameters: Glucose (non-fasting), Blood Urea Nitrogen (BUN), Creatinine, Sodium, Potassium, Calcium, Direct Bilirubin and Total Bilirubin (milligrams per decilitre) | Up to 3 months
Absolute values of Aspartate aminotransferase/serum glutamic-oxaloacetic transaminase, Alanine aminotransferase/serum glutamic-pyruvic transaminase, Alkaline phosphatase, Creatine phosphokinase (International Units per litre) | Up to 3 months
Absolute value of routine urinalysis: potential of hydrogen (pH) | Up to 3 months
Number of participants with abnormal urinalysis dipstick results: glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, leukocyte esterase | Up to 3 months
Change from baseline in haematology parameter: Platelet count (cells per microliter) | Baseline (Day 1) and up to 3 months
Change from baseline in haematology parameter: Red Blood Cell Count (RBC) (million cells per microliter) | Baseline (Day 1) and up to 3 months
Change from baseline in haematology parameter: Mean Corpuscle Volume (MCV) (Femtoliters) | Baseline (Day 1) and up to 3 months
Change from baseline in haematology parameter: Mean Corpuscle haemoglobin (MCH) (Picograms) | Baseline (Day 1) and up to 3 months
Change from baseline in haematology parameter: Reticulocytes (Percentage of reticulocytes) | Baseline (Day 1) and up to 3 months
Change from baseline in haematology parameters: Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils (giga cells per litre) | Baseline (Day 1) and up to 3 months
Change from baseline in haematology parameter: haemoglobin (Hgb) (grams per decilitre) | Baseline (Day 1) and up to 3 months
Change from baseline in haematology parameters: haematocrit (Proportion of red blood cells in blood) | Baseline (Day 1) and up to 3 months
Change from baseline in Clinical Chemistry parameters: Glucose (non-fasting), Blood Urea Nitrogen (BUN), Creatinine, Sodium, Potassium, Calcium, Direct Bilirubin and Total Bilirubin (milligrams per decilitre) | Baseline (Day 1) and up to 3 months
Change from baseline in Aspartate aminotransferase/ serum glutamic-oxaloacetic transaminase,Alanine aminotransferase/serum glutamic-pyruvic transaminase, Alkaline phosphatase, Creatine phosphokinase (International Units per litre) | Baseline (Day 1) and up to 3 months
Change from baseline in routine urinalysis: pH | Baseline (Day 1) and up to 3 months
Absolute values for vital signs: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) [millimeters of mercury (mm Hg)] | Up to 3 months
Absolute values for vital sign: pulse rate [beats per min (bpm)] | Up to 3 months
Change from baseline in vital signs: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) [millimeters of mercury (mm Hg)] | Baseline (Day 1) and up to 3 months
Change from baseline in vital sign: pulse rate [beats per min (bpm)] | Baseline (Day 1) and up to 3 months
Absolute values for 12 Lead Electrocardiograms (ECGs) in Corrected QT interval (QTc) (milliseconds) | Up to 3 months
Absolute values for heart rate [beats per min (bpm)] | Up to 3 months
Change from baseline for 12 Lead ECGs in QTc (milliseconds) | Baseline (Day 1) and up to 3 months
Change from baseline for heart rate [beats per min (bpm)] | Baseline (Day 1) and up to 3 months
Change from baseline in Asthma Control Questionnaire (ACQ-6) score | Baseline (Day 1) and up to 3 months
  ACQ-6 consists of 5 symptom related questions (nocturnal awakening, symptoms on waking in the morning, activity limitation, shortness of breath and wheeze with response options ranging from zero (no impairment/limitation) to 6 (total impairment/ limitation)) and a question on rescue bronchodilator use. A score of less than or equal to (<=) 0.75 indicates well-controlled asthma and a score greater than or equal to (>=)1.5 indicates poorly controlled asthma.
Change from baseline for pre-bronchodilator Forced expiratory volume in 1 second (FEV1) | Baseline (Day 1) and up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (94):
- United States (36):
  - GSK Investigational Site, North Hollywood, California
  - GSK Investigational Site, San Mateo, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Naples, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Winter Park, Florida
  - GSK Investigational Site, Rincon, Georgia
  - GSK Investigational Site, Stonecrest, Georgia
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Owensboro, Kentucky
  - GSK Investigational Site, Fall River, Massachusetts
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Minneota, Minnesota
  - GSK Investigational Site, Olive Branch, Mississippi
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Jersey City, New Jersey
  - GSK Investigational Site, Riverdale, New Jersey
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Dublin, Ohio
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Pottstown, Pennsylvania
  - GSK Investigational Site, Rock Hill, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Sugar Land, Texas
  - GSK Investigational Site, Tomball, Texas
- Argentina (3):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, La Plata
  - GSK Investigational Site, Mendoza
- Australia (4):
  - GSK Investigational Site, Botany, New South Wales
  - GSK Investigational Site, Coffs Harbour, New South Wales
  - GSK Investigational Site, Kanwal, New South Wales
  - GSK Investigational Site, Spearwood, Western Australia
- Canada (6):
  - GSK Investigational Site, Ajax, Ontario
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Québec, Quebec
- France (7):
  - GSK Investigational Site, Amiens
  - GSK Investigational Site, Argenteuil
  - GSK Investigational Site, Cannes
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Poitiers
  - GSK Investigational Site, Pontoise
  - GSK Investigational Site, Strasbourg
- Greece (3):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Larissa
  - GSK Investigational Site, Thessaloniki
- Italy (10):
  - GSK Investigational Site, Cagliari
  - GSK Investigational Site, Florence
  - GSK Investigational Site, Foggia
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Napoli
  - GSK Investigational Site, Padua
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Torino
  - GSK Investigational Site, Tradate VA
  - GSK Investigational Site, Verona
- GSK Investigational Site, Panama City, Panama
- GSK Investigational Site, Iloilo City, Philippines
- Poland (8):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Bielsko-Biala
  - GSK Investigational Site, Chorzów
  - GSK Investigational Site, Elblag
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Ostrowiec Świętokrzyski
  - GSK Investigational Site, Płock
  - GSK Investigational Site, Tarnów
- Spain (6):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Benalmádena
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marbella
  - GSK Investigational Site, Pozuelo de AlarcOn Madr
  - GSK Investigational Site, Santiago de Compostela
- GSK Investigational Site, Pathum Thani, Thailand
- United Kingdom (8):
  - GSK Investigational Site, Bebington
  - GSK Investigational Site, Cambridgeshire
  - GSK Investigational Site, Corby
  - GSK Investigational Site, Greater Manchester
  - GSK Investigational Site, Guisborough
  - GSK Investigational Site, Hounslow
  - GSK Investigational Site, Rhyl
  - GSK Investigational Site, Uttoxeter

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/